CLINICAL TRIAL: NCT02448966
Title: Traditional Three-incision Esophagectomy Versus Minimally Invasive Thorascopic/Laparoscopic Esophagectomy for cT1b-3N0-1M0 Thoracic Esophageal Cancer
Brief Title: Traditional Three-incision Esophagectomy Versus Minimally Invasive Thorascopic and Laparoscopic Esophagectomy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Collaborators: Peking University Cancer Hospital & Institute (Other); Henan Cancer Hospital (Other Government); Hebei Medical University Fourth Hospital (Other); Shanghai Zhongshan Hospital (Other); Harbin Medical University (Other); Sichuan Cancer Hospital and Research Institute (Other); Fujian Cancer Hospital (Other Government); Liaoning Cancer Hospital & Institute (Other); Hunan Cancer Hospital (Other); Sun Yat-sen University (Other); Zhejiang Cancer Hospital (Other); Tang-Du Hospital (Other); Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Jie He, President, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Other Study IDs: NKTRDP-2015BAI12B08-02
Record Dates: First submitted 2015-05-08; First posted 2015-05-20 (Estimated); Last update posted 2015-05-20 (Estimated); Status verified 2015-05

CONDITIONS: Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Traditional open esophagectomy: Treated by traditional three-incision esophagectomy in the centers with enough experience in esophagectomy via right thoracotomy and the volume ≧50 cases each year.
  Interventions: Procedure: open esophagectomy
- Minimally invasive eophagectomy: treated by minimally invasive thorascopic/laparoscopic esophagectomy in the centers with enough experience in VATS esophagectomy and the volume≧50 cases each year.
  Interventions: Procedure: Minimally invasive esophagectomy

INTERVENTIONS:
Procedure: open esophagectomy
  Groups: Traditional open esophagectomy
Procedure: Minimally invasive esophagectomy
  Groups: Minimally invasive eophagectomy

SUMMARY:
Esophageal carcinoma is an aggressive malignancy with poor prognosis. Surgical resection remains the most effective method for this malignant disease. VATS esophagectomy has become more and more popular in China and around the world. Although VATS esophagectomy has been proven to be effective in preventing respiratory complications, there is still no ample evidences to demonstrate that VATS esophagectomy is as effective as traditional three-incision esophagectomy in lymph node dissection and is equal or superior in long-term survival. The purpose of this large scale prospective observational study is to compare the minimally invasive thorascopic/laparoscopic esophagectomy with traditional three-incision esophagectomy in lymph node dissection, postoperative recovery, postoperative complications, and long-term survival.

DETAILED DESCRIPTION:
Esophageal carcinoma is an aggressive malignancy with poor prognosis,For these patients, radical esophagectomy is the cornerstone of multimodality treatment with curative intent. Transthoracic esophagectomy is the preferred surgical approach worldwide allowing for en-bloc resection of the tumor. However, the percentage of cardiopulmonary complications associated with the traditional three-incision esophagectomy is high.Recent studies have shown that the minimally invasive thorascopic and laparoscopic esophagectomy is at least equivalent to the open transthoracic approach for esophageal cancer in terms of short-term oncological outcomes,including reduced blood loss, shorter ICU stay,and lower pulmonary complication rate, but the evidence is not ample because the sample size is not enough.The objective of this study is to compare the efficacy, perioperative complications, lymph node dissection and long term survival between the thoracic esophageal cancer patients treated by minimally invasive thorascopic/laparoscopic esophagectomy and open transthoracic esophagectomy by three incisions.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically proven squamous cell esophageal cancer, without any previous anti-tumor therapy;
2. Preoperative clinical TNM stage:cT1b-3N0-1M0;
3. Adequate cardiopulmonary, liver, brain and kidney function which can tolerate the esophagectomy either via traditional tree-incision or minimally invasive thorascopic/laparoscopic esophagectomy;
4. Preoperative assessment by CT and EUS is fit for minimally invasive thorascopic/laparoscopic esophagectomy;
5. Willing to participate the clinical trial and sign the informed consent before being enrolled into clinical trail.

Exclusion Criteria:

1. Previous use of anti-cancer therapy;
2. Preoperative clinical TNM stage: N2-3 or M1;
3. Inadequate cardiopulmonary,liver, brain and kidney function for surgery;
4. Previous malignancy history;
5. Unwilling to participate the clinical trial and refuse to sign informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: cT1b-3N0-1M0 thoracic esophageal cancer.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2015-01; Primary Completion 2017-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Long term survival | 5 years

SECONDARY OUTCOMES:
Disease free survival | 5 years
Postoperative complications | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Jie He, MD,PhD, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China